CLINICAL TRIAL: NCT00602953
Title: Role of Pancreatic Triglyceride Content in Beta-cell Function
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ildiko Lingvay, MD, MPH, MSCS, University of Texas Southwestern Medical Center
Other Study IDs: 042007-021; 1K23RR02447001
Record Dates: First submitted 2007-10-25; First posted 2008-01-28 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Healthy volunteers: Normal weight and normal glucose tolerance.
  Interventions: Other: No intervention planned.
- Pre-diabetes: Impaired fasting glucose of impaired glucose tolerance.
  Interventions: Other: No intervention planned.
- Overweight: Overweight or obese volunteers, but with normal fasting and postprandial glucose levels.
  Interventions: Other: No intervention planned.
- Type 2 diabetes: Patients with type 2 diabetes.
  Interventions: Other: No intervention planned.
- Type 1 diabetes: Patients with type 1 diabetes.
  Interventions: Other: No intervention planned.

INTERVENTIONS:
Other: No intervention planned. — This is a cross-sectional observational study, no intervention is planned.

SUMMARY:
The study evaluates if fat accumulates in the pancreas in individuals at risk of developing obesity-related diabetes. It also evaluates if the amount of fat in the pancreas can predict the residual functional capacity of the pancreas (insulin secretion).

ELIGIBILITY:
Inclusion Criteria:

* adults without prior history of pancreatic disease (other than diabetes)

Exclusion Criteria:

* use of unapproved medications
* contraindications to the MRI procedure
* contraindications to frequent blood draws
* pregnancy
* use of more than 2 alcoholic drinks/day

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We enroll adult volunteers of all ethnicities who have no contraindications to the study procedures or use medications that interfere with our measurements.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2007-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ildiko Lingvay, MD, MPH, MSCS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Volunteers | Pre-diabetes | Overweight | Type 2 Diabetes | Type 1 Diabetes
Started | 15 | 26 | 47 | 13 | 0
Completed | 15 | 26 | 47 | 13 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Pre-diabetes | Overweight | Type 2 Diabetes | Type 1 Diabetes | Total
Number analyzed (Participants) | 15 | 26 | 47 | 13 | 0 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 26 | 47 | 13 | 0 | 101
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (8) | 41 (10) | 39 (9) | 47 (9) |  | 40 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 35 | 10 | 0 | 71
  Male | 4 | 11 | 12 | 3 | 0 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 26 | 47 | 13 |  | 101

OUTCOME MEASURES:

1. Primary Outcome: Pancreatic and Liver Fat
Description: Pancreatic and liver triglyceride (fat) content measured by the magnetic resonance spectroscopy (MRS) technique in volunteers with a wide range of body mass index (BMI).
Time Frame: Within 1 month after screening visit.
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Healthy Volunteers | Pre-diabetes | Overweight | Type 2 Diabetes | Type 1 Diabetes
Number analyzed (Participants) | 15 | 26 | 47 | 13 | 0
percent
  Pancreatic fat MRS | 1.87 [0.2 to 6.26] | 6.57 [1.90 to 17.93] | 3.61 [0.79 to 8.98] | 5.85 [3.43 to 13.96] |
  Liver fat MRS | 0.96 [0.61 to 1.83] | 4.09 [1.86 to 12.43] | 3.33 [1.29 to 6.99] | 8.76 [4.93 to 21.18] |

2. Primary Outcome: Beta-cell Function; AIRg - Acute Insulin Response to Glucose
Description: Beta-cell function as measured by frequently sampled intravenous glucose tolerance test (FSIVGTT) in volunteers with a wide range of body mass index (BMI).
  AIRg - acute insulin response to glucose. Blood samples were collected at -5, -1, 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 25, 30, 40, 50, 70, 100, 140, and 180 minutes, where time 0 is when an i.v. bolus of 50% glucose solution (0.3 g/kg) was injected.
Time Frame: At screening visit.
Measure: Median (Inter-Quartile Range); unit: microU/mL x min
Arm/Group | Healthy Volunteers | Pre-diabetes | Overweight | Type 2 Diabetes | Type 1 Diabetes
Number analyzed (Participants) | 15 | 26 | 47 | 13 | 0
microU/mL x min | 197.55 [118.15 to 237.42] | 321.09 [151.71 to 446.46] | 519.33 [385.59 to 927.69] | 8.9 [1.0 to 56.58] |

3. Primary Outcome: Insulin Sensitivity (SI)
Description: Sensitivity index measured during frequently sampled intravenous glucose tolerance test (FSIVGTT) in volunteers with a wide range of body mass index (BMI).
  Blood samples were collected at -5, -1, 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 25, 30, 40, 50, 70, 100, 140, and 180 minutes, where time 0 is when an i.v. bolus of 50% glucose solution (0.3 g/kg) was injected. Higher numbers indicates better insulin sensitivity Insulin sensitivity was estimated as Matsuda index using formula = 10,000 / (FPG x FPI x Glucosemean0-180 x Insulinmean0-180)0.5, where FPG = fasting plasma glucose and FPI = fasting plasma insulin.
Time Frame: At screening visit.
Measure: Median (Inter-Quartile Range); unit: min-1 per pU/mL x 10v4
Arm/Group | Healthy Volunteers | Pre-diabetes | Overweight | Type 2 Diabetes | Type 1 Diabetes
Number analyzed (Participants) | 15 | 26 | 47 | 13 | 0
min-1 per pU/mL x 10v4 | 5.48 [3.85 to 7.46] | 2.28 [1.6 to 4.55] | 2.29 [1.54 to 2.84] | 1.55 [1.28 to 3.76] |

4. Primary Outcome: Disposition Index (DI)
Description: Disposition index measured during frequently sampled intravenous glucose tolerance test (FSIVGTT) in volunteers with a wide range of body mass index (BMI). Blood samples were collected at -5, -1, 2, 3, 4, 5, 6, 8, 10, 14, 19, 22, 25, 30, 40, 50, 70, 100, 140, and 180 minutes, where time 0 is when an i.v. bolus of 50% glucose solution (0.3 g/kg) was injected. Disposition index (DI) was used to characterize the correlation between β-cell sensitivity and insulin sensitivity and was determined using formula DI = AIRg x SI (from outcomes 2 and 3). Higher numbers indicates a better improvement in beta-cell function.
Time Frame: At screening visit.
Measure: Median (Inter-Quartile Range); unit: Number
Arm/Group | Healthy Volunteers | Pre-diabetes | Overweight | Type 2 Diabetes | Type 1 Diabetes
Number analyzed (Participants) | 15 | 26 | 47 | 13 | 0
Number | 1001.8 [744.52 to 1332.1] | 739.84 [478.15 to 1026.53] | 1031.26 [749.6 to 1796.35] | 15.61 [4.31 to 133.19] |

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Healthy Volunteers | Pre-diabetes | Overweight | Type 2 Diabetes | Type 1 Diabetes
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/26 | 0/47 | 0/13 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/26 | 0/47 | 0/13 | 0/0
Other Adverse Events (participants affected / at risk) | 0/15 | 0/26 | 0/47 | 0/13 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No